CLINICAL TRIAL: NCT01441505
Title: A Study of Ketamine as an Antidepressant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Collaborators: Wesley Mission (Other)
Responsible Party: Principal Investigator, Colleen Loo, Associate Professor, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HREC 10409
Record Dates: First submitted 2011-09-16; First posted 2011-09-27 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — Ketamine; Sodium Chloride; Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ketamine — Ketamine IV, IM, or SC will be administered in Phase I and II
Drug: Saline or Midazolam (active placebo) — Saline, or midazolam 0.01mg/kg will be administered in Phase I

SUMMARY:
Recently, interest has emerged in the use of ketamine as an antidepressant. Recent placebo-controlled clinical trials administering a single dose and an open label trial giving repeated doses shown that ketamine is markedly superior to placebo at reducing depression, including in treatment-resistant patients, and that its antidepressant effects have a very rapid onset.

This clinical study consists of two phases. In Phase I, participants who satisfy inclusion criteria will receive ketamine at variable doses (0.1mg/kg-0.5mg/kg) or a placebo (saline, or 0.01mg/kg midazolam) once a week over up to 6 weeks. If participants qualify for Phase II, they will receive repeated sessions of ketamine at variable doses over three weeks. During both phases, mood, psychiatric, and neuropsychological outcomes will be measured.

DETAILED DESCRIPTION:
This clinical study consists of two phases. In Phase I, participants will receive variable doses of intravenous, intramuscular, or subcutaneous ketamine (0.1-0.5mg/kg) or placebo (saline, or 0.01mg/kg midazolam) weekly for up to 6 consecutive weeks. Prior to receiving ketamine/placebo, participants' mood and psychiatric symptoms will be assessed. Once they have received their treatment, mood, psychiatric side effects, ketamine blood levels, heart rate, blood pressure and biomarkers will be assessed. Mood and cognitive performance be assessed again after 4 hours. Finally, mood will also be assessed the next day.

Some participants may be eligible to continue to Phase II. In this phase, participants will receive doses of ketamine approximately weekly for up to 6 months. During this phase, participants' mood, psychiatric, biomarkers and cognitive outcomes will be assessed.

The purpose of the trial is to investigate the antidepressant and safety effects of using ketamine as a treatment in depression.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV-TR criteria for Major Depressive Episode
* 18 years or over
* Able to give informed consent

Exclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, rapid cycling bipolar disorder, or current psychotic symptoms
* Known sensitivity or contraindication to ketamine
* Recent drug abuse
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on depression rating scales | Before, 4 hours after, and 24 hours after ketamine session

SECONDARY OUTCOMES:
Psychiatric side effects (BPRS, CADSS) and memory tests | Cognitive battery done before and after 3 weeks; side effects measured immediately before and 4 hours after each ketamine session in both phases.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K Loo, MB BS FRANZCP MD, Principal Investigator — University of New South Wales
Locations (1):
- Wesley Hospital, Kogarah, New South Wales, Australia

REFERENCES:
- [Background] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Background] Larkin GL, Beautrais AL. A preliminary naturalistic study of low-dose ketamine for depression and suicide ideation in the emergency department. Int J Neuropsychopharmacol. 2011 Sep;14(8):1127-31. doi: 10.1017/S1461145711000629. Epub 2011 May 5. PMID 21557878 (Retraction: PMID 28637184 Int J Neuropsychopharmacol. 2017 Jul 1;20(7):611)
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Derived] George D, Galvez V, Martin D, Kumar D, Leyden J, Hadzi-Pavlovic D, Harper S, Brodaty H, Glue P, Taylor R, Mitchell PB, Loo CK. Pilot Randomized Controlled Trial of Titrated Subcutaneous Ketamine in Older Patients with Treatment-Resistant Depression. Am J Geriatr Psychiatry. 2017 Nov;25(11):1199-1209. doi: 10.1016/j.jagp.2017.06.007. Epub 2017 Jun 13. PMID 28739263
- [Derived] Loo CK, Galvez V, O'Keefe E, Mitchell PB, Hadzi-Pavlovic D, Leyden J, Harper S, Somogyi AA, Lai R, Weickert CS, Glue P. Placebo-controlled pilot trial testing dose titration and intravenous, intramuscular and subcutaneous routes for ketamine in depression. Acta Psychiatr Scand. 2016 Jul;134(1):48-56. doi: 10.1111/acps.12572. Epub 2016 Mar 30. PMID 27028832
- See also: Related Info — http://www.blackdoginstitute.org.au